## Examining the Efficacy of a Tri-Compartment Unloader Knee Brace During Physical Rehabilitation in Non-Surgical Patients with Anterior Knee Pain

Statistical Analysis Plan
NCT05428332
June 28, 2022

Differences in baseline characteristics (age, gender, race, marital status, and laterality) between the brace and control groups were analyzed using Mann-Whitney U-tests and Fisher's exact tests due to small sample sizes and non-normally distributed continuous variables. Normality was assessed visually using histograms. Differences in patient reported outcome measures between the brace and control groups at baseline, 6-week follow-up, and 3-month follow-up were analyzed using Mann-Whitney U-tests and Fisher's exact tests. For each of the EQ-5D dimensions, responses were categorized into "no problem" and "any problem" (combining slight, moderate, severe, and extreme problems). Rates of experiencing "any problem" were analyzed between groups. Analyses were completed in RStudio using a two-sided level of significance of 0.05.